CLINICAL TRIAL: NCT01139346
Title: Phase I Study of Oral Darinaparsin in Advanced Solid Tumors
Brief Title: Study of Oral Darinaparsin in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGC1004
Record Dates: First submitted 2010-06-04; First posted 2010-06-08 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Advanced Solid Tumors
Keywords: carcinoma; sarcoma; metastatic; solid tumor
MeSH Terms: conditions — Carcinoma; Sarcoma; Neoplasm Metastasis | interventions — darinaparsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- oral darinaparsin (Experimental): open label, single arm, dose escalation
  Interventions: Drug: darinaparsin

INTERVENTIONS:
Drug: darinaparsin — dose escalating, starting at 200 mg twice per day for 21 days continuous followed by a 7 day rest per cycle.
  Other Names: ZIO-101-C; S-dimethylarsino-glutathione; Zinapar (TM)

SUMMARY:
This study is a Phase I, dose escalation study of oral darinaparsin for the treatment of advanced solid tumors. Eligible patients could have received any amount of previous therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histological or cytological confirmation of advanced cancer (solid tumor) that is refractory to standard therapies for their condition;
* Men and women of ≥18 years of age;
* ECOG performance score ≤2
* Eligible subjects with solid tumors MUST have at least one measurable lesion as defined by RECIST 1.1 guidelines. If the measurable disease is restricted to a solitary lesion, its neoplastic nature should be confirmed by cytology/histology. Measurable lesions MUST NOT have been in a previously irradiated field or injected with biological agents;
* Life expectancy ≥12 weeks;
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements, to be conducted <2 weeks prior to Baseline:

  * Creatinine ≤1.5 × upper limit of normal (ULN) OR a calculated creatinine clearance ≥50 cc/min
  * Total bilirubin ≤2 × ULN
  * Alanine transaminase (ALT) and aspartate transaminase (AST)≤3 × ULN
  * Granulocytes in peripheral blood ≥1 × 109/L, hemoglobin ≥10 g/dL, and platelets ≥50,000 /µL
* Adequate vascular access for repeated blood sampling;
* Men and women of childbearing potential must agree to use effective contraception from Screening through the duration of Study participation;
* Written informed consent in compliance with ZIOPHARM policies and the Human Investigation Review Committee (IEC/IRB) having jurisdiction over the site.

Exclusion Criteria:

* Arsenic allergy.
* New York Heart Association (NYHA) functional class ≥3 myocardial infarction (see Appendix 3) within 6 months.
* Uncontrolled cardiac arrhythmia other than asymptomatic atrial fibrillation; a QTc ≥450 msec; or a ≥Grade 2 atrioventricular (AV) block or left bundle branch block (LBBB); or documented history of prolonged QTc.
* Pregnant and/or lactating women.
* Uncontrolled systemic infection (documented with microbiological studies).
* Metastatic brain or meningeal tumors.
* Patients with seizure disorder requiring medication (such as anti-epileptics)
* History of confusion or dementia or neurological condition that could mask a potential adverse response to the Study Drug, which may include transient ischemic attack, Parkinson's disease, thrombotic or hemorrhagic stroke, Alzheimer's, and other neurological disorders.
* Anticancer chemotherapy or immunotherapy during the study or within four weeks of Study entry (mitomycin C or nitrosureas should not be given within 6 weeks of Study entry)
* Radiotherapy during study or within 3 weeks of Study entry.
* Major surgery within 4 weeks of start of Study Drug dosing.
* Other Investigational drug therapy during this trial within four weeks prior to Study entry.
* History of invasive second primary malignancy diagnosed within the previous 3 years except for Stage I endometrial/cervical carcinoma or prostate carcinoma treated surgically, and non-melanoma skin cancer.
* Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of Study results.
* Any condition that is unstable or could jeopardize the safety of the patient and his/her compliance in the Study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Determine Toxicity Profile | One Year
  a primary outcome measure is to determine the toxicity profile of oral darinaparsin when given continuously for 21 days followed by a 7 day rest period per cycle
Determine Maximum Tolerated Dose | One Year
  a primary outcome measure is to determine the maximum tolerated dose of oral darinaparsin when given continuously for 21 days followed by a 7 day rest period per cycle
Determine the preliminary activity/efficacy | One Year
  a primary outcome measure is to determine the preliminary activity/efficacy of oral darinaparsin when given continuously for 21 days followed by a 7 day rest period per cycle
Determine Pharmacokinetic profile | One Year
  a primary outcome measure is to determine the pharmacokinetic profile of oral darinaparsin when given continuously for 21 days followed by a 7 day rest period per cycle

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan J. Lewis, MD, PhD, Study Director — ZIOPHARM, Oncology, Inc.
Locations (3):
- United States (3):
  - Lafayette, Indiana
  - Dallas, Texas
  - Houston, Texas